CLINICAL TRIAL: NCT04179994
Title: Comparison of Clinical Efficacy of a Miswak Extract-Containing Toothpaste to a Dentifrice Containing Potassium Nitrate and to a Placebo on Dentinal Hypersensitivity: A Randomized Clinical Trial
Brief Title: Efficacy of Miswak Extract Toothpaste as Compared Potassium Nitrate in The Management of Dentinal Hypersensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Abdulrahman Alshehri, Principal Investigator, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MoHSaudiArabia
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: The study will be a single-center, longitudinal, triple-masked (for participants, operators, and statistician), equal ratio, randomized non-crossover design.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Miswak extract-containing toothpaste group (Experimental): Test group.
  Interventions: Other: Miswak extract-containing toothpaste
- Toothpaste containing Potassium Nitrates (Active Comparator): Positive control.
  Interventions: Other: Potassium nitrates-containing toothpaste
- Placebo group (Placebo Comparator): Toothpaste contains same ingredients of test group except for the active ingredient as negative control.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Miswak extract-containing toothpaste — Miswak extract-containing toothpaste will be applied to the tooth diagnosed with DH
  Other Names: Test group
  Arms: Miswak extract-containing toothpaste group
Other: Potassium nitrates-containing toothpaste — Potassium nitrates-containing toothpaste will be applied to the tooth diagnosed with DH
  Other Names: Positive control
  Arms: Toothpaste containing Potassium Nitrates
Other: Placebo — A toothpaste containing the same ingredients of the test toothpaste except for the active ingredient
  Other Names: Negative control as placebo
  Arms: Placebo group

SUMMARY:
The study will be a single-center, longitudinal, triple-masked (for participants, operators, and statistician), equal ratio, randomized non-crossover design. The study designed following the criteria described by Holland et al 1997. The current experiments will follow CONSORT guidelines and will be registered at the US National Institutes of Health (ClinicalTrials.gov). The sensitivity scores will be measured at three intervals: at baseline, at 2 weeks, and at 6 weeks. The duration of the current study estimated to be 6 weeks and will be conducted between January 2020 and March 2020. The study protocol will be submitted initially to the Ethical Committee of the Aseer Central Hospital, Aseer region, Saudi Arabia. After getting the approval and facilitation letters, the participants will be selected randomly from patients attending periodontal clinics at Aseer Dental Center, Aseer region.

DETAILED DESCRIPTION:
Three toothpastes will be investigated during the study period that are 1) commercially available miswak extract-containing toothpaste; 2) commercially available toothpaste containing 5% potassium nitrate as positive control; 3) a toothpaste containing the same formulation as miswak extract except for the active ingredient (miswak extract) as negative control. Toothpastes will be dispensed in labeled containers named A,B, and C to achieve the triple masking for investigators, participants, and statisticians. Masked toothpastes will be revealed to the investigators after the statistical analyses.

After allocation, all subjects will be instructed to refrain from using any desensitizing agents for two weeks prior to the study up to the end of study period. The randomization process will be made using SPSS, the function "RAND" to assign every subject to random A, B, or C masked toothpastes. Moreover, to insure the blinded process of the study we will dispense the toothpastes in a previously prepared similar containers in separate area. Two trained examiners will read and record the scores each visit (baseline, 2-weeks, and 6-weeks). For the seek of examiners' calibration, Kappa statistic will be used to assess the inter-rater reproducibility and we will duplicate a 10% of the study results.

During each visit, teeth around the targeted tooth will be isolated with cotton rolls then the stimuli will be applied using a sharp dental explorer. It will be passed across the facial area of the tooth, perpendicular to the tooth long axis. The average of three consecutive applications will be recorded as a the reading for that tooth.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with history of DH caused by cervical erosion or gingival recession
* Subjects show good general health
* Must have at least two teeth with VAS score of 4 or more

Exclusion Criteria:

* Subjects have teeth with caries, occlusal restorations, or orthodontic appliances
* Subjects allergic to ingredients used in the study
* Subjects present any oral pathology, eating disorders, chronic disease, or any disease requiring repeated or regular analgesia, anti-inflammatory drugs, or antihistamines

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-04-25 (Estimated); Study Completion 2020-07-25 (Estimated)

PRIMARY OUTCOMES:
Pain reduction | 6 weeks period
  Visual Analog Scale (VAS) will be used to measure pain intensity. The scale is graded from 1 to 10 with zero score indicates a pain-free response and 10 indicates sever pain or discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Alshehri, MS, Principal Investigator — Ministry of Health, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
We can share these data for the seek of spreading knowledge in any case if there is no conflicts for any body.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From June 2020 to January 2021.
Access Criteria: Data can be send to a researchers who will get scientific benefit of them. By mean of paper or electronic mails.

REFERENCES:
- [Background] Al-Otaibi M, Al-Harthy M, Gustafsson A, Johansson A, Claesson R, Angmar-Mansson B. Subgingival plaque microbiota in Saudi Arabians after use of miswak chewing stick and toothbrush. J Clin Periodontol. 2004 Dec;31(12):1048-53. doi: 10.1111/j.1600-051X.2004.00618.x. PMID 15560804
- [Background] BRAENNSTROEM M, ASTROEM A. A STUDY ON THE MECHANISM OF PAIN ELICITED FROM THE DENTIN. J Dent Res. 1964 Jul-Aug;43:619-25. doi: 10.1177/00220345640430041601. No abstract available. PMID 14183350
- [Background] Canadian Advisory Board on Dentin Hypersensitivity. Consensus-based recommendations for the diagnosis and management of dentin hypersensitivity. J Can Dent Assoc. 2003 Apr;69(4):221-6. PMID 12662460
- [Background] Cunha-Cruz J, Wataha JC, Heaton LJ, Rothen M, Sobieraj M, Scott J, Berg J; Northwest Practice-based Research Collaborative in Evidence-based DENTistry. The prevalence of dentin hypersensitivity in general dental practices in the northwest United States. J Am Dent Assoc. 2013 Mar;144(3):288-96. doi: 10.14219/jada.archive.2013.0116. PMID 23449905
- [Background] Douglas-de-Oliveira DW, Vitor GP, Silveira JO, Martins CC, Costa FO, Cota LOM. Effect of dentin hypersensitivity treatment on oral health related quality of life - A systematic review and meta-analysis. J Dent. 2018 Apr;71:1-8. doi: 10.1016/j.jdent.2017.12.007. Epub 2017 Dec 17. PMID 29262305
- [Background] Dowell P, Addy M. Dentine hypersensitivity--a review. Aetiology, symptoms and theories of pain production. J Clin Periodontol. 1983 Jul;10(4):341-50. doi: 10.1111/j.1600-051x.1983.tb01283.x. PMID 6309917
- [Background] Favaro Zeola L, Soares PV, Cunha-Cruz J. Prevalence of dentin hypersensitivity: Systematic review and meta-analysis. J Dent. 2019 Feb;81:1-6. doi: 10.1016/j.jdent.2018.12.015. Epub 2019 Jan 11. PMID 30639724
- [Background] Gillam DG, Seo HS, Bulman JS, Newman HN. Perceptions of dentine hypersensitivity in a general practice population. J Oral Rehabil. 1999 Sep;26(9):710-4. doi: 10.1046/j.1365-2842.1999.00436.x. PMID 10520145
- [Background] Hattab FN. Meswak: the natural toothbrush. J Clin Dent. 1997;8(5):125-9. PMID 9487831
- [Background] Holland GR, Narhi MN, Addy M, Gangarosa L, Orchardson R. Guidelines for the design and conduct of clinical trials on dentine hypersensitivity. J Clin Periodontol. 1997 Nov;24(11):808-13. doi: 10.1111/j.1600-051x.1997.tb01194.x. PMID 9402502
- [Background] Markowitz K, Kim S. The role of selected cations in the desensitization of intradental nerves. Proc Finn Dent Soc. 1992;88 Suppl 1:39-54. PMID 1508896
- [Background] Rees JS, Addy M. A cross-sectional study of buccal cervical sensitivity in UK general dental practice and a summary review of prevalence studies. Int J Dent Hyg. 2004 May;2(2):64-9. doi: 10.1111/j.1601-5029.2004.00068.x. PMID 16451464
- [Background] Schiff T, Dotson M, Cohen S, De Vizio W, McCool J, Volpe A. Efficacy of a dentifrice containing potassium nitrate, soluble pyrophosphate, PVM/MA copolymer, and sodium fluoride on dentinal hypersensitivity: a twelve-week clinical study. J Clin Dent. 1994;5 Spec No:87-92. PMID 8534380
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Sofrata A, Santangelo EM, Azeem M, Borg-Karlson AK, Gustafsson A, Putsep K. Benzyl isothiocyanate, a major component from the roots of Salvadora persica is highly active against Gram-negative bacteria. PLoS One. 2011;6(8):e23045. doi: 10.1371/journal.pone.0023045. Epub 2011 Aug 1. PMID 21829688
- [Background] Vongsavan N, Matthews B. Fluid flow through cat dentine in vivo. Arch Oral Biol. 1992 Mar;37(3):175-85. doi: 10.1016/0003-9969(92)90087-o. PMID 1586280
- [Background] West NX. Dentine hypersensitivity: preventive and therapeutic approaches to treatment. Periodontol 2000. 2008;48:31-41. doi: 10.1111/j.1600-0757.2008.00262.x. No abstract available. PMID 18715354
- [Background] Yoshiyama M, Noiri Y, Ozaki K, Uchida A, Ishikawa Y, Ishida H. Transmission electron microscopic characterization of hypersensitive human radicular dentin. J Dent Res. 1990 Jun;69(6):1293-7. doi: 10.1177/00220345900690061401. PMID 2355124
- [Result] Azaripour A, Mahmoodi B, Habibi E, Willershausen I, Schmidtmann I, Willershausen B. Effectiveness of a miswak extract-containing toothpaste on gingival inflammation: a randomized clinical trial. Int J Dent Hyg. 2017 Aug;15(3):195-202. doi: 10.1111/idh.12195. Epub 2015 Dec 22. PMID 26694786
- [Result] Dragolich WE, Pashley DH, Brennan WA, O'Neal RB, Horner JA, Van Dyke TE. An in vitro study of dentinal tubule occlusion by ferric oxalate. J Periodontol. 1993 Nov;64(11):1045-51. doi: 10.1902/jop.1993.64.11.1045. PMID 8295089
- [Result] Gallob J, Sufi F, Amini P, Siddiqi M, Mason S. A randomised exploratory clinical evaluation of dentifrices used as controls in dentinal hypersensitivity studies. J Dent. 2017 Sep;64:80-87. doi: 10.1016/j.jdent.2017.06.009. Epub 2017 Jun 23. PMID 28652142
- [Result] Gupta P, Agarwal N, Anup N, Manujunath BC, Bhalla A. Evaluating the anti-plaque efficacy of meswak (Salvadora persica) containing dentifrice: A triple blind controlled trial. J Pharm Bioallied Sci. 2012 Oct;4(4):282-5. doi: 10.4103/0975-7406.103238. PMID 23248560
- [Result] Mason S, Kingston R, Shneyer L, Harding M. Clinical study to monitor dentinal hypersensitivity with episodic use of a desensitising dentifrice. BDJ Open. 2017 Jun 23;3:17011. doi: 10.1038/bdjopen.2017.11. eCollection 2017. PMID 29789771
- [Result] Pradeep AR, Sharma A. Comparison of clinical efficacy of a dentifrice containing calcium sodium phosphosilicate to a dentifrice containing potassium nitrate and to a placebo on dentinal hypersensitivity: a randomized clinical trial. J Periodontol. 2010 Aug;81(8):1167-73. doi: 10.1902/jop.2010.100056. PMID 20370417